CLINICAL TRIAL: NCT04128696
Title: A Randomized, Double-blind, Adaptive, Phase II/III Study of GSK3359609 or Placebo in Combination With Pembrolizumab for First-Line Treatment of PD-L1 Positive Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Study of GSK3359609 and Pembrolizumab in Programmed Death Receptor 1-ligand 1 (PD-L1) Positive Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Acronym: INDUCE-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was stopped by the sponsor based on assessment of the clinical data
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 209229; 2019-002263-99 (EudraCT Number)
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Neoplasms, Head and Neck
Keywords: GSK3359609; Pembrolizumab; Programmed death receptor 1-ligand 1; Head and neck squamous cell carcinoma/cancer; Inducible T cell co-stimulatory receptor; Keynote-A01; Head & neck; Phase III
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This will be a randomized, parallel group treatment study with eligible participants receiving GSK3359609 plus pembrolizumab or placebo plus pembrolizumab.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving feladilimab and pembrolizumab (Experimental): Participants were administered feladilimab (humanized anti-ICOS immunoglobulin G4 [IgG4] monoclonal antibody [mAb]) and pembrolizumab (humanized anti-PD-1 IgG4 mAb) as an intravenous (IV) infusion once every three weeks.
  Interventions: Drug: feladilimab; Drug: Pembrolizumab
- Participants receiving placebo and pembrolizumab (Active Comparator): Participants were administered placebo and pembrolizumab (humanized anti-PD-1 IgG4 mAb) as an IV infusion once every three weeks.
  Interventions: Drug: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: feladilimab — feladilimab is available as an intravenous infusion.
  Arms: Participants receiving feladilimab and pembrolizumab
Drug: Pembrolizumab — Pembrolizumab is available as an intravenous infusion.
Drug: Placebo — Placebo is available as an intravenous infusion.
  Arms: Participants receiving placebo and pembrolizumab

SUMMARY:
The purpose of study is to evaluate if the addition of GSK3359609 to pembrolizumab as first-line treatment improves the efficacy of pembrolizumab in participants with recurrent or metastatic (R/M) head and neck squamous cell carcinoma/cancer (HNSCC).This is a randomized, double-blind, adaptive Phase II/III study comparing a combination of GSK3359609 inducible T cell co-stimulatory receptor (ICOS) agonist and pembrolizumab to pembrolizumab plus placebo in participants with programmed death receptor 1-ligand 1 (PD-L1) combined positive score (CPS) >=1 R/M HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent
* Male or female, age >=18 years
* Histological or cytological documentation of Head and Neck Squamous Cell Carcinoma (HNSCC) that is considered incurable by local therapies
* Primary tumor location of the oral cavity, oropharynx, hypopharynx or larynx
* No prior systemic therapy administered in the recurrent or metastatic setting (except for systemic therapy given as part of multimodal treatment for locally advanced disease)
* Measurable disease per RECIST version 1.1 guidelines
* ECOG Performance PS score of 0 or 1
* Adequate organ function
* Life expectancy of at least 12 weeks
* Female participants: must not be pregnant, not breastfeeding, and at least one of the following conditions apply:

  1. Not a woman of childbearing potential (WOCBP)
  2. A WOCBP who agrees to use a method of birth control from 30 days prior to randomization and for at least 120 days after the last dose of study treatment
* Male participants with female partners of child-bearing potential: must agree to use a highly effective contraception while receiving study treatment and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period
* Provide tumor tissue from excisional or core biopsy (fine needle aspirates and bone biopsies are not acceptable) acquired within 2 years prior to randomization for PD-L1 immunohistochemistry (IHC) testing by central laboratory
* Have PD-L1 Immunohistochemistry (IHC) CPS 1 status by central laboratory testing
* Have results from testing of Human Papilloma Virus (HPV) status for oropharyngeal cancer

Exclusion Criteria:

* Prior therapy with an anti-PD-1/L1/L2 and/or anti-ICOS directed agent
* Systemic approved or investigational anticancer therapy within 30 days or 5 half-lives of the drug, whichever is shorter
* Major surgery 28 days prior to randomization
* Has high risk of bleeding
* Toxicity related to prior treatment that has not resolved to <=Grade 1 (except alopecia, hearing loss, endocrinopathy managed with replacement therapy, and peripheral neuropathy which must be<= Grade 2)
* Received transfusion of blood products or administration of colony stimulating factors within 14 days prior to randomization
* Central nervous system (CNS) metastases, with the following exception: Participants with asymptomatic CNS metastases who are clinically stable and have no requirement for steroids for at least 14 days prior to randomization
* Invasive malignancy or history of invasive malignancy other than disease under study within the last 3 years, except as noted below:

  a. Any other invasive malignancy for which the participant was definitively treated, has been disease-free for 3 years and in the opinion of the principal investigator and GSK Medical Monitor will not affect the evaluation of the effects of the study treatment on the currently targeted malignancy, may be included in this clinical study
* Autoimmune disease or syndrome that required systemic treatment within the past 2 years
* Has a diagnosis of immunodeficiency or is receiving systemic steroids (≥10 mg oral prednisone per day or equivalent) or other immunosuppressive agents within 7 days prior to randomization
* Receipt of any live vaccine within 30 days prior randomization
* Prior allogeneic/autologous bone marrow or solid organ transplantation
* Has current pneumonitis or history of non-infectious pneumonitis that required steroids or other immunosuppressive agents
* Recent history (within the past 6 months) of uncontrolled symptomatic ascites, pleural or pericardial effusions
* Recent history (within the past 6 months) of gastrointestinal obstruction that required surgery, acute diverticulitis, inflammatory bowel disease, or intra-abdominal abscess
* Recent history of allergen desensitization therapy within 4 weeks of randomization
* History or evidence of cardiac abnormalities within the 6 months prior to randomization
* Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice
* Active infection requiring systemic therapy
* Known HIV infection, or positive test for hepatitis B active infection (presence of hepatitis B surface antigen), or hepatitis C active infection
* History of severe hypersensitivity to monoclonal antibodies or any ingredient used in the study treatment formulations
* Known history of active tuberculosis
* Any serious and/or unstable pre-existing medical (aside from malignancy), psychiatric disorder, or other condition that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures in the opinion of the investigator
* Is currently participating in (unless in follow-up phase and 4 weeks have elapsed from last dose of prior investigational agent), or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to date of randomization
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (145):
- United States (13):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Seattle, Washington
- Argentina (4):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, San Juan
- Australia (7):
  - GSK Investigational Site, Blacktown, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Darlinghurst
- Brazil (6):
  - GSK Investigational Site, Vitória, Espírito Santo
  - GSK Investigational Site, Florianópolis, Santa Catarina
  - GSK Investigational Site, Barretos, São Paulo
  - GSK Investigational Site, São José do Rio Preto, São Paulo
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, São Paulo
- Canada (8):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Rimouski, Quebec
- China (10):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanning, Guangxi
  - GSK Investigational Site, Guiyang, Guizhou
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Nanchang, Jiangxi
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Bengbu
  - GSK Investigational Site, Harbin
  - GSK Investigational Site, Hefei
  - GSK Investigational Site, Shnghai
- GSK Investigational Site, Copenhagen, Denmark
- France (10):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Epagny Metz-Tessy
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Valenciennes
- Germany (5):
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (2):
  - GSK Investigational Site, Heraklion,Crete
  - GSK Investigational Site, Thessaloniki
- GSK Investigational Site, Dublin, Ireland
- Israel (3):
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
- Italy (5):
  - GSK Investigational Site, Meldola (FC), Emilia-Romagna
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Candiolo, Piedmont
  - GSK Investigational Site, Legnago (VR), Veneto
- Japan (15):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Mexico (2):
  - GSK Investigational Site, Saltillo, Coahuila
  - GSK Investigational Site, Guadalajara, Jalisco
- Netherlands (2):
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
- Norway (2):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
- Poland (7):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Gliwice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Tomaszów Mazowiecki
  - GSK Investigational Site, Warsaw
- Portugal (4):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Matosinhos Municipality
  - GSK Investigational Site, Porto
- Romania (11):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Floreşti
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Otopeni
  - GSK Investigational Site, Satu Mare
  - GSK Investigational Site, Suceava
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Poselok Kuzmolovsky
  - GSK Investigational Site, Pushkin
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yaroslavl
- South Korea (5):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Hwasun,Jeollanam-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Switzerland (2):
  - GSK Investigational Site, Sankt Gallen
  - GSK Investigational Site, Zurich
- Taiwan (4):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan
- United Kingdom (4):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a data sharing agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 315 participants with recurrent or metastatic head and neck squamous cell carcinoma/cancer (HNSCC) were enrolled in this study.
Pre-assignment Details: Recruitment in the study was stopped following review of interim safety and efficacy data by the Independent Data Monitoring Committee, after a pre-specified futility analysis. A Dear Investigator Letter (DIL) was issued to stop screening/randomization of further subjects to the study.
Groups:
- Participants Receiving Feladilimab and Pembrolizumab: Participants were administered feladilimab (GSK3359609-humanized anti-ICOS immunoglobulin G4 [IgG4] monoclonal antibody [mAb]) and pembrolizumab (humanized anti-PD-1 IgG4 mAb) as an intravenous (IV) infusion once every three weeks (Q3W).
- Participants Receiving Placebo and Pembrolizumab: Participants were administered placebo and pembrolizumab (humanized anti-PD-1 IgG4 mAb) as an IV infusion Q3W.
Period: Overall Study
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Started (Enrolled population) | 158 | 157
Modified Intent to Treat (mITT) Population (2 participants (1 from each arm) were dosed after the date of DIL requesting immediate discontinuation of feladilimab/placebo and were not included in the mITT population.) | 157 | 156
Safety Population (Two participants were initially randomized to placebo+pembrolizumab arm but were dosed with feladilimab. Therefore, they were included in the in the feladilimab+pembrolizumab arm of the safety population. The 2 participants enrolled but excluded from the mITT population (one from each arm) were both included in the placebo+pembrolizumab arm for the safety population, as both participants were only dosed with pembrolizumab.) | 159 | 156
Completed | 115 | 98
Not Completed | 43 | 59
Not completed — Lost to Follow-up | 3 | 7
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Study Closed/Terminated | 26 | 38
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Participants Receiving Feladilimab and Pembrolizumab: Participants were administered feladilimab (GSK3359609-humanized anti-ICOS IgG4 mAb) and pembrolizumab (humanized anti-PD-1 IgG4 mAb) as an IV infusion Q3W.
- Total: Total of all reporting groups
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab | Total
Number analyzed (Participants) | 158 | 157 | 315
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 95 | 79 | 174
  ≥65-84 years | 62 | 76 | 138
  ≥85 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 129 | 126 | 255
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 2 | 0 | 2
  Asian - East Asian Heritage | 19 | 22 | 41
  Asian - Japanese Heritage | 12 | 7 | 19
  Black or African American | 4 | 2 | 6
  Missing | 3 | 6 | 9
  Mixed White Race | 1 | 1 | 2
  Multiple | 1 | 0 | 1
  White - Arabic/North African Heritage | 4 | 1 | 5
  White - White/Caucasian/European Heritage | 111 | 118 | 229
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in the Programmed Death Receptor-ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1 Population
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells. Kaplan-Meier estimate for the median OS is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 16 months
Population: mITT: All randomized participants, whether or not randomized intervention was administered, excluding those who were first dosed or randomized after the date of DIL requesting immediate discontinuation of feladilimab /placebo. This analysis was based on the study intervention to which the participant was randomized. All participants with PD-L1 CPS ≥1 in the mITT population were analyzed.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 157 | 156
Week | 44.1 [35.9 to NA] — The upper limit of the 95% CI was not calculable from the available data at the time of data cut off. | NA [52.4 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; The hazard ratio and 2-sided 95% CI was calculated from the Cox regression model with Efron's method of tie handling, a treatment covariate and stratified by PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20) and HPV status (oropharynx HPV positive vs oropharynx HPV negative/unknown and non-oropharynx); Test type: Superiority; p = 0.973, Stratified Cox proportional hazard model — Nominal p-value was calculated based on the one-sided log-rank test, stratified by PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20) and HPV status (oropharynx HPV positive vs oropharynx HPV negative/unknown and non-oropharynx); Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.99 to 2.29]

2. Primary Outcome: OS in the PD-L1 Expression High (CPS ≥20) Population
Description: as for outcome 1
Time Frame: Up to approximately 16 months
Population: Data for participants with PD-L1 CPS ≥20 in mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 70 | 69
Week | 42.1 [25.4 to NA] — The upper limit of the 95% CI was not calculable from the available data at the time of data cut off. | NA [52.4 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; The hazard ratio and 2-sided 95% CI was calculated from the Cox regression model with Efron's method of tie handling, a treatment covariate and stratified by HPV status (oropharynx HPV positive vs oropharynx HPV negative/unknown and non-oropharynx); Test type: Superiority; p > 0.999, Stratified Cox proportional hazard model — Nominal p-value was calculated based on the one-sided log-rank test, stratified by HPV status (oropharynx HPV positive vs oropharynx HPV negative/unknown and non-oropharynx); Hazard Ratio (HR) = 4.44, 95% CI 2-sided [2.01 to 9.82]

3. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) in the PD-L1 CPS ≥1 Population
Description: PFS per RECIST version (v)1.1 was defined as the time from the date of randomization to the date of first documented disease progression or death due to any cause, whichever occurs first. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells. Kaplan-Meier estimate for the median PFS is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 16 months
Population: All participants with PD-L1 CPS ≥1 in the mITT population were analyzed.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 157 | 156
Week | 10.1 [9.1 to 15.0] | 16.0 [14.3 to 26.1]
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.989, Stratified Cox proportional hazard model — Nominal p-value was calculated based on the log-rank test, stratified by stratified by PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20) and HPV status (oropharynx HPV positive vs oropharynx HPV negative/unknown and non-oropharynx); Hazard Ratio (HR) = 1.40, 95% CI 2-sided [1.05 to 1.86]

4. Secondary Outcome: PFS Per Immune-based RECIST (iRECIST) in the PD-L1 CPS ≥1 Population
Description: PFS per iRECIST was defined as the interval of time from the date of randomization to the date of the first documented disease progression confirmed consecutively per iRECIST based on investigator assessment, or death due to any cause, whichever occurs first. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells. Kaplan-Meier estimate for the median PFS is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 16 months
Population: All participants with PD-L1 CPS ≥1 in the mITT population were analyzed.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 157 | 156
Week | 13.0 [9.1 to 15.1] | 21.4 [15.6 to 27.0]
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.996, Stratified Cox proportional hazard model — Nominal p-value was calculated based on the log-rank test, stratified by PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20) and HPV status (oropharynx HPV positive vs oropharynx HPV negative/unknown and non-oropharynx); Hazard Ratio (HR) = 1.48, 95% CI 2-sided [1.10 to 1.99]

5. Secondary Outcome: PFS Per RECIST in the PD-L1 CPS ≥20 Population
Description: PFS per RECIST v1.1 was defined as the time from the date of randomization to the date of first documented disease progression per RECIST v1.1. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells. Kaplan-Meier estimate for the median PFS is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method.
Time Frame: Up to approximately 16 months
Population: Data for participants with PD-L1 CPS ≥20 in mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 70 | 69
Week | 13.0 [8.6 to 26.1] | 21.1 [15.6 to 32.9]
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Stratified Cox proportional hazard model; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [0.98 to 2.43]

6. Secondary Outcome: PFS Per iRECIST (iPFS) in the PD-L1 CPS ≥20 Population
Description: as for outcome 4
Time Frame: Up to approximately 16 months
Population: Data for participants with PD-L1 CPS ≥20 in mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 70 | 69
Week | 13.1 [8.6 to 26.7] | 26.7 [20.1 to 32.9]
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Stratified Cox proportional hazard model; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [1.00 to 2.53]

7. Secondary Outcome: Milestone OS Rate at 12 Months in the PD-L1 CPS ≥1 Population
Description: Milestone OS rate at 12 months was estimated using the Kaplan-Meier method. Associated 95% confidence intervals are estimated using the Brookmeyer-Crowley method. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: 12 months
Population: All participants with PD-L1 CPS ≥1 in the mITT population were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 157 | 156
Percentage of participants | 44.0 [30.0 to 58.0] | 68.0 [57.0 to 77.0]

8. Secondary Outcome: Milestone OS Rate at 24 Months in the PD-L1 CPS ≥1 Population
Description: Milestone OS rate at 24 months was not evaluated. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: 24 months
Population: All participants with PD-L1 CPS ≥1 in the mITT population were to be analyzed. Data for this endpoint were not collected as all participants were on the study for < 24 months, the maximum duration of follow-up was approximately 16 months.
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Milestone OS Rate at 12 Months in the PD-L1 CPS ≥20 Population
Description: as for outcome 7
Time Frame: 12 months
Population: Data for participants with PD-L1 CPS ≥20 in mITT population are presented.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 70 | 69
Percentage of participants | 46.0 [28.0 to 63.0] | 88.0 [76.0 to 94.0]

10. Secondary Outcome: Milestone OS Rate at 24 Months in the PD-L1 CPS ≥20 Population
Description: as for outcome 8
Time Frame: 24 months
Population: Participants with PD-L1 CPS ≥20 in the mITT population were to be analyzed. Data for this endpoint were not collected as all participants were on the study for <24 months, the maximum duration of follow-up was approximately 16 months.
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Overall Response Rate (ORR) Per RECIST v1.1 in the PD-L1 CPS ≥1 Population
Description: ORR per RECIST v1.1 was defined as the proportion of the participants who have a complete response (CR) or partial response (PR) as the best overall response per RECIST v1.1 based upon investigator assessment. As a randomized double-blind study in which primary endpoints are OS and PFS, the confirmation of CR and PR was not required. Rate and associated 2-sided 95 percent Exact (Clopper-Pearson) Confidence Intervals are provided for each treatment arm which are unadjusted. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 16 months
Population: All participants with PD-L1 CPS ≥1 in the mITT population were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 157 | 156
Percentage of Participants | 19.7 [13.8 to 26.8] | 25.0 [18.4 to 32.6]
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; The comparison between the treatment groups was based on the stratified Miettinen & Nurminen method with strata weighting by sample size and a single treatment covariate. Stratification factors included PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20) and HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Other; Difference in Percentage = -5.3, 95% CI 2-sided [-14.6 to 4.0]

12. Secondary Outcome: ORR Per RECIST v1.1 in the PD-L1 CPS ≥20 Population
Description: ORR per RECIST v1.1 was defined as the proportion of the participants who have a CR or PR as the best overall response per RECIST v1.1 based upon investigator assessment. As a randomized double-blind study in which primary endpoints are OS and PFS, the confirmation of CR and PR was not required. Rate and associated 2-sided 95 percent Exact (Clopper-Pearson) Confidence Intervals are provided for each treatment arm which are unadjusted. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 16 months
Population: Data for participants with PD-L1 CPS ≥20 in mITT population are presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 70 | 69
Percentage of Participants | 20.0 [11.4 to 31.3] | 33.3 [22.4 to 45.7]
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; The comparison between the treatment groups was based on the stratified Miettinen & Nurminen method with strata weighting by sample size and a single treatment covariate. Stratification factors included HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Other; Difference in Percentage = -13.3, 95% CI 2-sided [-27.8 to 1.5]

13. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1 in the PD-L1 CPS ≥1 Population
Description: DCR per RECIST v1.1 based upon investigator assessment, was defined as the percentage of participants with a best overall response of CR or PR at any time plus stable disease (SD) meeting the minimum time of 15 weeks. A status of SD≥15 weeks will be assigned if the follow-up disease assessment has met the SD criteria at least once after the date of randomization at a minimum of 14 weeks (98 days) considering a one-week visit window. Rate and associated 2-sided 95 percent Exact (Clopper-Pearson) Confidence Intervals are provided for each treatment arm which are unadjusted. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 16 months
Population: All participants with PD-L1 CPS ≥1 in the mITT population were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 157 | 156
Percentage of Participants | 33.1 [25.8 to 41.1] | 44.9 [36.9 to 53.0]
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; The comparison between treatment groups was based on the stratified Miettinen & Nurminen method with strata weighting by sample size and a single treatment covariate. Stratification factors included PD-L1 expression (CPS ≥20 vs. 1≤ CPS <20) and HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Other; Difference in Percentage = -11.8, 95% CI 2-sided [-22.4 to -1.1]

14. Secondary Outcome: DCR Per RECIST v1.1 in the PD-L1 CPS ≥20 Population
Description: as for outcome 13
Time Frame: Up to approximately 16 months
Population: Data for participants with PD-L1 CPS ≥20 in mITT population are presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 70 | 69
Percentage of Participants | 37.1 [25.9 to 49.5] | 55.1 [42.6 to 67.1]
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; The comparison between treatment groups was based on the stratified Miettinen & Nurminen method with strata weighting by sample size and a single treatment covariate. Stratification factors included HPV status (positive vs. negative). Participants with oropharynx HPV negative/unknown and non-oropharyngeal tumors were combined as the HPV negative group; Test type: Other; Difference in Percentage = -18.0, 95% CI 2-sided [-33.7 to -1.4]

15. Secondary Outcome: Duration of Response (DoR) Per RECIST v1.1 in the PD-L1 CPS ≥1 Population
Description: DoR per RECIST v1.1 is defined as the time from first documented evidence of CR or PR until first documented disease progression per RECIST v1.1 based upon investigator assessment or death due to any cause, whichever occurs first, among participants who demonstrated CR or PR as the best overall response per RECIST v1.1. Kaplan-Meier estimate for the median DoR is presented, along with associated 95% confidence interval, estimated using the Brookmeyer-Crowley method. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 16 months
Population: Data for participants with a best overall response of CR or PR in the mITT population with PD-L1 CPS ≥1 are presented.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 31 | 39
Weeks | NA [NA to NA] — The median was not reached at the time of data cut off. The upper and lower limit of the 95% CI was not calculable from the available data at the time of data cut off. | NA [20.6 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.

16. Secondary Outcome: DoR Per RECIST v1.1 in the PD-L1 CPS ≥20 Population
Description: as for outcome 15
Time Frame: Up to approximately 16 months
Population: Data for participants with a best overall response of CR or PR in the mITT population with PD-L1 CPS ≥20 are presented.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 14 | 23
Weeks | NA [18.1 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off. | NA [12.1 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.

17. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, any other situation such as important medical events according to medical or scientific judgement.
Time Frame: Up to approximately 43 months
Population: Safety Population: All randomized participants who take at least 1 dose of study intervention. Participants were assigned to the actual study intervention group of feladilimab + pembrolizumab if the participant received any dose of feladilimab. Participants were analyzed according to the actual study intervention received.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 159 | 156
Participants
  Any AE | 150 | 145
  Any SAE | 52 | 53

18. Secondary Outcome: Number of Participants With AEs by Severity
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity of each AE was reported during the study and was assigned a grade according to the National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE). AEs severity were graded on a 5-point scale as: 1 = mild; discomfort noticed, but no disruption to daily activity, 2 = moderate; discomfort sufficient to reduce or affect normal daily activity, 3 = severe; inability to work or perform normal daily activity, 4 = life-threatening consequences and 5 = death related to AE.
Time Frame: Up to approximately 43 months
Population: Safety Population: All randomized participants who take at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 159 | 156
Participants
  Grade 1 | 34 | 21
  Grade 2 | 48 | 54
  Grade 3 | 46 | 46
  Grade 4 | 7 | 6
  Grade 5 | 15 | 18

19. Secondary Outcome: Number of Participants With SAEs by Severity
Description: An SAE was defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, any other situation such as important medical events according to medical or scientific judgement. Severity of each SAE was reported during the study and was assigned a grade according to the NCI-CTCAE. SAEs severity were graded on a 5-point scale as: 1 = mild; discomfort noticed, but no disruption to daily activity, 2 = moderate; discomfort sufficient to reduce or affect normal daily activity, 3 = severe; inability to work or perform normal daily activity, 4 = life-threatening consequences and 5 = death related to AE. Data of participants experiencing SAEs of Grade ≥3 have been presented.
Time Frame: Up to approximately 43 months
Population: Safety Population: All randomized participants who take at least 1 dose of study intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 159 | 156
Participants | 43 | 46

20. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: AESI were defined as events of potential immunologic etiology, including immune-related AEs (irAEs). Such events recently reported after treatment with other immune modulatory therapy include colitis, uveitis, hepatitis, pneumonitis, diarrhea, endocrine disorders, and specific cutaneous toxicities, as well as other events that may be immune mediated.
Time Frame: Up to approximately 43 months
Population: All participants in the safety population were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 159 | 156
Participants | 49 | 67

21. Secondary Outcome: Number of Participants With AESI by Severity
Description: AESI were defined as events of potential immunologic etiology, including immune-related AEs (irAEs). Such events recently reported after treatment with other immune modulatory therapy include colitis, uveitis, hepatitis, pneumonitis, diarrhea, endocrine disorders, and specific cutaneous toxicities, as well as other events that may be immune mediated. Severity of each AESI was reported during the study and was assigned a grade according to the NCI-CTCAE. AESIs severity were graded on a 5-point scale as: 1 = mild; discomfort noticed, but no disruption to daily activity, 2 = moderate; discomfort sufficient to reduce or affect normal daily activity, 3 = severe; inability to work or perform normal daily activity, 4 = life-threatening consequences and 5 = death related to AE. Data of participants experiencing AESIs of Grade ≥3 have been presented.
Time Frame: Up to approximately 43 months
Population: All participants in the safety population were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 159 | 156
Participants | 2 | 6

22. Secondary Outcome: Number of Participants With Dose Modifications
Description: Number of participants with dose modifications (including dose interruptions, dose delays and treatment discontinuations) were reported by each interventional component.
Time Frame: Up to approximately 16 months
Population: All participants in the safety population were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 159 | 156
Participants
  Dose interruption by component - feladilimab | 4 | NA — Participants in this treatment arm were not dosed with feladilimab
  Dose interruption by component - placebo | NA — Participants in this treatment arm were not dosed with placebo | 1
  Dose interruption by component - pembrolizumab | 0 | 1
  Dose delays by component - feladilimab | 9 | NA — Participants in this treatment arm were not dosed with feladilimab
  Dose delays by component - placebo | NA — Participants in this treatment arm were not dosed with placebo | 5
  Dose delays by component - pembrolizumab | 11 | 6
  Treatment discontinuation by component - feladilimab/placebo | 159 | 154
  Treatment discontinuation by component - pembrolizumab | 108 | 93

23. Secondary Outcome: Time to Deterioration (TTD) in Pain in the PD-L1 CPS ≥1 Population
Description: TTD in pain is defined as the time from randomization to the first definitive meaningful deterioration from baseline in the European Organization for Research and Treatment of Cancer Item Library(EORTC IL51) pain domain, i.e. an increase from baseline of at least 8.33 observed at all subsequent non-missing visits. The EORTC Quality of Life Questionnaire 35-Item Head and Neck Module (QLQ-H&N35) is a head and neck specific module with multi-item scales. The questionnaire scores for each scale and single-item measure are averaged and transformed linearly to present a score ranging from 0-100. A high score represents a high/healthy level of functioning. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 16 months
Population: All participants with PD-L1 CPS ≥1 in the mITT population were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 157 | 156
Months | 6.3 [5.1 to NA] — The upper limit of the 95% CI was not calculable from the available data at the time of data cut off. | 10.4 [6.3 to NA] — The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.783, Stratified Cox proportional hazard model — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.78 to 1.77]

24. Secondary Outcome: TTD in Pain in the PD-L1 CPS ≥20 Population
Description: TTD in pain is defined as the time from randomization to the first definitive meaningful deterioration from baseline in the EORTC IL51 pain domain, i.e. an increase from baseline of at least 8.33 observed at all subsequent non-missing visits. The EORTC QLQ-H&N35 is a head and neck specific module with multi-item scales. The mouth pain, swallowing, speech problems, opening mouth, coughing, feeding tube, and trouble with social eating domains were administered and referred to as the EORTC IL51. The questionnaire scores for each scale and single-item measure are averaged and transformed linearly to present a score ranging from 0-100. A high score represents a high/healthy level of functioning. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 16 months
Population: Data for participants with PD-L1 CPS ≥20 in mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 70 | 69
Months | NA [5.1 to NA] — The median was not reached at the time of data cut off. The upper limit of the 95% CI was not calculable from the available data at the time of data cut off. | 12 [6.3 to NA] — The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.500, Stratified Cox proportional hazard model — Nominal p-value was calculated based on the log-rank test, stratified by HPV status (oropharynx HPV positive vs oropharynx HPV negative/unknown and non-oropharynx); Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.50 to 2.00]

25. Secondary Outcome: TTD in Physical Function in the PD-L1 CPS ≥1 Population
Description: TTD in physical function is defined as the time from randomization to the first definitive meaningful deterioration from baseline in the PF T-score, i.e. a decrease from baseline of at least 2.4 observed at all subsequent non-missing visits, as measured by the PROMIS PF 8c. The PROMIS PF 8c is an 8-item fixed length short form derived from the PROMIS Physical Function item bank. It includes a 5-point scale with three sets of response options. Scores on the PROMIS PF 8c are reported on a T score metric (mean = 50 and SD = 10), with higher scores reflecting better physical functioning. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 16 months
Population: All participants with PD-L1 CPS ≥1 in the mITT population were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 157 | 156
Months | 4.9 [3.5 to 7.7] | 4.9 [3.0 to 6.3]
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.329, Stratified Cox proportional hazard model — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.62 to 1.34]

26. Secondary Outcome: TTD in Physical Function in the PD-L1 CPS ≥20 Population
Description: TTD in physical function is defined as the time from randomization to the first definitive meaningful deterioration from baseline in the PF T-score, i.e. a decrease from baseline of at least 2.4 observed at all subsequent non-missing visits, as measured by the PROMIS PF 8c. The PROMIS PF 8c is an 8-item fixed length short form derived from the PROMIS Physical Function item bank. It includes a 5-point scale with three sets of response options. Scores on the PROMIS PF 8c are reported on a T score metric (mean = 50 and SD = 10), with higher scores reflecting better physical functioning. Data are presented for the PD-L1 CPS >=1 participants from mITT population. CPS was defined as the ratio of the combined number of PD-L1 expressing tumor cells and immune cells (lymphocytes and macrophages) to the total number of viable tumor cells.
Time Frame: Up to approximately 16 months
Population: Data for participants with PD-L1 CPS ≥20 in mITT population are presented.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
Number analyzed (Participants) | 70 | 69
Months | 4.9 [2.1 to NA] — The upper limit of the 95% CI was not calculable from the available data at the time of data cut off. | 4.9 [3.1 to NA] — The upper limit of the 95% CI was not calculable from the available data at the time of data cut off.
Statistical Analysis 1: Comparison: Participants Receiving Feladilimab and Pembrolizumab vs Participants Receiving Placebo and Pembrolizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.608, Stratified Cox proportional hazard model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.60 to 2.00]

ADVERSE EVENTS:
Time Frame: All cause mortality, non-SAEs and SAEs were collected from Day 1 to up to approximately 43 months.
Description: 2 participants were initially randomized to placebo+pembrolizumab arm but were dosed with feladilimab. Therefore, they were included in feladilimab+pembrolizumab arm of the safety population. The 2 participants enrolled but excluded from the mITT population (1 from each arm) were both included in placebo+pembrolizumab arm for the safety population, as both were only dosed with pembrolizumab.
Arm/Group | Participants Receiving Feladilimab and Pembrolizumab | Participants Receiving Placebo and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 116/159 | 97/156
Serious Adverse Events (participants affected / at risk) | 52/159 | 53/156
Other Adverse Events (participants affected / at risk) | 125/159 | 128/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Receiving Feladilimab and Pembrolizumab (N=159) | Participants Receiving Placebo and Pembrolizumab (N=156)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oral cavity fistula (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 4 (4)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (6) | 4 (4)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 2 (3) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Fistula discharge (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 6 (6)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Distributive shock (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 4 (5) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Receiving Feladilimab and Pembrolizumab (N=159) | Participants Receiving Placebo and Pembrolizumab (N=156)
Anaemia (Blood and lymphatic system disorders) | 26 (42) | 21 (26)
Hypothyroidism (Endocrine disorders) | 20 (20) | 16 (16)
Constipation (Gastrointestinal disorders) | 22 (28) | 24 (26)
Diarrhoea (Gastrointestinal disorders) | 21 (25) | 13 (19)
Dysphagia (Gastrointestinal disorders) | 17 (17) | 15 (15)
Nausea (Gastrointestinal disorders) | 17 (21) | 17 (20)
Vomiting (Gastrointestinal disorders) | 12 (15) | 8 (8)
Asthenia (General disorders) | 17 (17) | 14 (23)
Fatigue (General disorders) | 29 (30) | 29 (32)
Pyrexia (General disorders) | 11 (13) | 11 (12)
Alanine aminotransferase increased (Investigations) | 9 (10) | 12 (16)
Aspartate aminotransferase increased (Investigations) | 12 (15) | 11 (15)
Blood alkaline phosphatase increased (Investigations) | 8 (9) | 4 (4)
Weight decreased (Investigations) | 20 (20) | 27 (29)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15) | 28 (28)
Hypercalcaemia (Metabolism and nutrition disorders) | 11 (14) | 8 (10)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (17) | 7 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 13 (25) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (16) | 11 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 12 (12)
Headache (Nervous system disorders) | 15 (19) | 14 (17)
Insomnia (Psychiatric disorders) | 15 (15) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 11 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 19 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (15) | 17 (19)
Rash (Skin and subcutaneous tissue disorders) | 9 (12) | 21 (32)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 9 (11)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (9)
Anxiety (Psychiatric disorders) | 8 (8) | 3 (3)
COVID-19 (Infections and infestations) | 5 (5) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT04128696/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT04128696/SAP_001.pdf